## STATISTICAL ANALYSIS PLAN

Project Title: Perioperative pregabalin as part of a multimodal treatment plan for pain after

ureteroscopy with stent placement: a pilot

IRB Number: 2013680 Version Number: 1.1 Version Date: 11/20/2019

Principal Investigator: Katie Murray, DO

Funding Source: Departmental Clinical Trial Phase: Not Phased

Clinicaltrials.gov Number: NCT03927781 Study Drug/Study Device: Pregabalin

| Principal Investigator | Katie Murray, DO | Department of Surgery Urology |
|---|---|---|
| | | Division |
| Co-Investigator | Geoffrey Rosen, MD | Department of Surgery Urology Division |
| Consenting Professional(s) | Donartment of Surgery | DIVISION |
| Consenting Professional(s) | Department of Surgery- | |
| Department | Urology | |

University of Missouri University Hospital Department of Surgery Urology Division 1 Hospital Drive Columbia, MO 65212 Descriptive statistics (counts, proportions, medians) will be used to describe all data. We will describe the demographic information of the patients enrolled and the number of patients approached to meet full enrollment. We will assess the proportion who anticipated needing opioid pain medication, who appropriately received pregabalin, who received opioid pain medication at discharge, who had emergency room visits or hospitalizations in the first 30 post-operative days, and who received opioid prescriptions within the first 30 post-operative days. We will describe the number of oral morphine equivalents prescribed. We will include median USSQ scores. We will describe proportions reporting possible adverse effects and pain level reported. All analyses will be performed in R version 3.5.1. There will be no statistical tests performed.